CLINICAL TRIAL: NCT07293429
Title: Effects of Combined Posture Correction Exercise and Resistive Respiratory Muscle Training on Dyspnea, Chest Expansion, Craniovertebral Angle and Pulmonary Function Test, in COPD Patients With Forward Head Posture
Brief Title: Combined Posture Correction and Resistive Respiratory Muscles Training in COPD With FHP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kaynat saleem
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease; Forward Head Posture
Keywords: craniovertebral angle; resistive training; posture correction; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistive inspiratory muscles training (Experimental): GROUP A: will be treated with resistive inspiratory muscles training along with posture correction exercises
  Interventions: Device: Resistive inspiratory muscles training
- Resistive expiratory muscles training (Experimental): GROUP B: will be treated with Resistive expiratory muscles training along with posture correction exercises
  Interventions: Device: Resistive expiratory muscles training:
- Combined resistive inspiratory and expiratory muscles training (Experimental): GROUP C: will be treated with Combined resistive inspiratory and expiratory muscles training along with posture correction exercises
  Interventions: Device: Resistive inspiratory muscles training; Device: Combined resistive inspiratory and expiratory muscles training

INTERVENTIONS:
Device: Resistive inspiratory muscles training — Resistive Inspiratory Muscle Training (IMT) will be implemented using a threshold inspiratory muscle trainer, which requires patients to inhale through a one-way valve that provides adjustable resistance. The training sessions will begin with patients sitting comfortably in an upright position to optimize lung function. They will be instructed to take a deep breath, ensuring their diaphragm engages fully, and then inhale through the device, which will resist airflow, thereby increasing the workload on the inspiratory muscles. Initially, the resistance will be set at a level that is challenging yet achievable, with the aim to gradually increase resistance as the patient's strength and endurance improve. Each session will last 30 minutes, consisting of intervals of resisted inhalation followed by brief rest periods. Patients will perform 3 sets of 10 breaths with appropriate breaks in between. The training will be conducted 3 times per week,
  Arms: Combined resistive inspiratory and expiratory muscles training; Resistive inspiratory muscles training
Device: Resistive expiratory muscles training: — Resistive Expiratory Muscle Training (EMT) will be employed to enhance the strength and endurance of the expiratory muscles in COPD patients. This training will utilize a threshold expiratory muscle trainer, designed to provide resistance during exhalation, thereby engaging the abdominal and intercostal muscles effectively. Patients will begin each session in a comfortable, upright position to optimize lung function. They will be instructed to take a deep inhalation to fully expand their lungs, and then exhale forcefully through the device against the resistance. The resistance level will be adjustable and initially set to a manageable level, with plans to gradually increase it as the patient's strength improves. Each training session will last 30 minutes, consisting of intervals of resisted exhalation followed by brief recovery periods. Patients will perform 3 sets of 10 breaths, with appropriate breaks in between. it will be performed 3 times per week
  Arms: Resistive expiratory muscles training
Device: Combined resistive inspiratory and expiratory muscles training — Resistive Inspiratory and Expiratory Muscle Training will be implemented concurrently as a comprehensive approach to enhance the strength and endurance of both inspiratory and expiratory muscles in COPD patients. During each session, patients will utilize a threshold inspiratory muscle trainer for inhalation while simultaneously using a threshold expiratory muscle trainer for exhalation. Each training session will last 20-30 minutes, beginning with patients taking a deep breath to fully engage their diaphragm before inhaling through the inspiratory trainer and exhaling forcefully against the resistance of the expiratory trainer. Patients will perform 3 sets of 10 breaths, with appropriate breaks in between to prevent fatigue and ensure effective training. This resistive EMT protocol will be conducted 3 times per week
  Arms: Combined resistive inspiratory and expiratory muscles training

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by persistent respiratory symptoms and airflow limitation, often exacerbated by postural abnormalities such as forward head posture (FHP). FHP can lead to significant alterations in breathing patterns, reducing the efficiency of respiratory muscles and impairing lung function. Patients with COPD and FHP frequently exhibit muscular imbalances, where overactive accessory muscles compensate for weakened primary respiratory muscles Resistive Inspiratory Muscle Training strengthens inhalation muscles using resistance devices to enhance respiratory function in COPD patients. Resistive Expiratory Muscle Training focuses on strengthening exhalation muscles through resistance during exhalation, improving breathing efficiency. Posture Correction Exercises address forward head posture by stretching tight muscles and strengthening weak ones to optimize breathing mechanics. Combined Resistive Inspiratory and Expiratory Muscle Training integrates both inspiratory and expiratory muscle training, using resistance for both inhalation and exhalation, to maximize respiratory efficiency and overall lung function in COPD patients. The objective of the study is to determine the effects of combined exercise and resistive respiratory muscles training on dyspnea, chest expansion, craniovertebral angle and pulmonary function test, in COPD patients with forward head posture.

Patients of COPD with forward head posture will be recruited by convenient sampling technique using seal opaque method. 72 patients will be equally divided into three groups with 24 patients each. Posture correction exercises will be added as baseline treatment for all three groups session. GROUP A will be treated with resistive inspiratory muscles training (RIMT). GROUP B will be treated with resistive expiratory muscles training (REMT). GROUP C will be treated with combined resistive inspiratory and expiratory muscles technique (RIMT+REMT).treatment session will be of 8 weeks and will include three reading (pre, post treatment and one follow-up). Outcomes measurement will include; dyspnea by dyspnea 12 questionnaires, chest expansion by measuring tape, craniovertebral angle by radiograph and pulmonary function test by spirometer. Data will be analyzed by SPSS software version 21.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of COPD at stage 1 and 2

  * COPD with forward head posture.
  * Craniovertebral angle < 53 degrees (20)
  * Age 40-60
  * Both genders
  * Spirometric evidence of significant chronic air-flow limitation (ie, FEV1 of 50% of predicted and FEV1/FVC ratio of 70% of predicted) in whom COPD had been diagnosed (21)
  * Persistent dyspnea with a self-rated intensity of ⩾6 (out of 10) on a visual analogue
  * Having muscular tightness (pectoralis major and minor, upper trapezius, sternocleidomastoid)

Exclusion Criteria:

* • COPD with severe complications (respiratory infections, acute exacerbations, pulmonary hypertension)

  * COPD with cardiovascular complications (Cor Pulmonale, atherosclerosis, risk of venous thromboembolism)
  * Unstable respiratory, neurological, and cardiovascular conditions
  * Congenital Cervical/spinal deformity
  * Patients with frozen shoulder, shoulder, cervical radiculopathy)
  * Uncontrolled underlying conditions(22)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Dyspnea-12 questionnaire: | pretreatment, 4th week, 8th week
  The Dyspnoea-12 (D-12), particularly evaluates both the physical and emotional components of dyspnea, was created to provide a quick, reliable assessment that is applicable to a wide range of cardiorespiratory conditions. Twelve items on the D-12 measure dyspnea on a four-point scale from none to mild, moderate, and severe. The physical domain is the sum of the scores for the first seven items, which range from 0 to 21. The affective domain scores, which range from 0 to 15, are the sum of the remaining five items. The D-12 total scores, which range from 0 to 36, are the sum of the twelve items. Severity can be determined by higher scores.
  The test provided significant evidence of assessing characteristics such as construct validity, internal consistency, and structural validity in the Norwegian-language D-12
Measuring tape | pretreatment, 4th week, 8th week
  The tape measure is a conventional instrument used to assess chest expansion. It measures circumferentially at predetermined spots on the chest wall. Assuring that the underlying soft tissues have not been compressed will assist in helping the tape conform to the chest wall. (24) A tape is used at two distinct rib cage positions to quantify chest expansion. Three anatomical landmarks for thoracic expansion will be the angle of Louis on sternum, xiphoid process of mid chest expansion, midpoint between the xiphoid process and umbilicus for lower chest expansion.
  Measurements of chest expansion performed with a tape on the upper and lower thoracic levels have a strong relationship and exhibit good intra- and inter-rater reliability and consistency.
Radiograph | pretreatment, 4th week, 8th week
  One of the common objective methods for evaluating head posture is the measurement of craniovertebral (CV) angle. It is the angle formed when a line drawn horizontally through the seventh cervical (C7) vertebra's spinous process and a line connecting it to the tragus of ear.
  Radiographic measurements play a crucial role in assessing cervical spine alignment in the sagittal plane by evaluating the relative positions of the vertebrae and joints
Spirometer | pretreatment, 4th week, 8th week
  A spirometer is a device that measures the amount of air that a person can inhale and exhale during a predetermined period of time. This measurement is typically performed to diagnose lung diseases, specifically blockage and reorganization, forced vital capacity (FVC), and forced expiratory volume in one second (FEV1) are a few spirometer characteristics that are utilized for clinical assessment. The existence or lack of anomalies in the lung can be detected using two of the three measures. Spirometry is an easy, safe, non-invasive, and reasonably priced diagnostic tool for identifying airflow blockage. Spirometry, one of the currently available methods for the early detection of asthma and COPD, is therefore very crucial. It is advised that patients with asthma and COPD measure their static and dynamic respiratory functions every day in order to easily monitor their lung health and avoid exacerbations.

SECONDARY OUTCOMES:
COPD assessment test (CAT) | pretreatment, 4th week, 8th week
  The COPD Assessment Test (CAT) will be used to evaluate the quality of life in all participants. It is expected to serve as a straightforward and effective tool for assessing the health status of Thai COPD patients. The CAT consists of eight questions that address various aspects of the disease, including dyspnea, cough, sputum production, wheezing, fatigue, sleep disturbances, limitations in daily activities, social life, emotional well-being, and a sense of control. The CAT score ranges from 0 to 40, with the following classifications: a score of <10 indicates a low impact on health status, 11-20 indicates a moderate impact, 21-30 indicates a high impact, and >30 indicates a very high impact on health status.

CONTACTS AND LOCATIONS:
Overall Officials: wajeeha zia, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garratt AM, Nerheim EM, Einvik G, Stavem K, Edvardsen A. Evaluation of the Norwegian version of the Dyspnoea-12 questionnaire in patients with COPD. BMJ Open Respir Res. 2022 May;9(1):e001262. doi: 10.1136/bmjresp-2022-001262. PMID 35609940
- [Background] Ray AD, Udhoji S, Mashtare TL, Fisher NM. A combined inspiratory and expiratory muscle training program improves respiratory muscle strength and fatigue in multiple sclerosis. Arch Phys Med Rehabil. 2013 Oct;94(10):1964-70. doi: 10.1016/j.apmr.2013.05.005. Epub 2013 May 25. PMID 23714277
- [Background] Vazquez-Gandullo E, Hidalgo-Molina A, Montoro-Ballesteros F, Morales-Gonzalez M, Munoz-Ramirez I, Arnedillo-Munoz A. Reply to Yigit, S.; Akinci, B. Comment on "Vazquez-Gandullo et al. Inspiratory Muscle Training in Patients with Chronic Obstructive Pulmonary Disease (COPD) as Part of a Respiratory Rehabilitation Program Implementation of Mechanical Devices: A Systematic Review. Int. J. Environ. Res. Public Health 2022, 19, 5564". Int J Environ Res Public Health. 2023 Mar 9;20(6):4801. doi: 10.3390/ijerph20064801. PMID 36981710
- [Background] Postma K, Haisma JA, Hopman MT, Bergen MP, Stam HJ, Bussmann JB. Resistive inspiratory muscle training in people with spinal cord injury during inpatient rehabilitation: a randomized controlled trial. Phys Ther. 2014 Dec;94(12):1709-19. doi: 10.2522/ptj.20140079. Epub 2014 Jul 31. PMID 25082923
- [Background] Morais N, Cruz J, Marques A. Posture and mobility of the upper body quadrant and pulmonary function in COPD: an exploratory study. Braz J Phys Ther. 2016 Jul-Aug;20(4):345-54. doi: 10.1590/bjpt-rbf.2014.0162. Epub 2016 Apr 8. PMID 27556391
- [Background] Gupta N, Agrawal S, Chakrabarti S, Ish P. COPD 2020 Guidelines - what is new and why? Adv Respir Med. 2020;88(1):38-40. doi: 10.5603/ARM.2020.0080. No abstract available. PMID 32153009